CLINICAL TRIAL: NCT02993380
Title: Effect of Cooked Olive Oil on Erythrocyte Membrane Fatty Acid Contents in Hemodialysis Patients
Brief Title: Effect of Olive Oil on Erythrocyte Membrane Fatty Acid Contents in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, WON SUK AN, Professor, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OliveHD_2016
Record Dates: First submitted 2016-12-09; First posted 2016-12-15 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Hemodialysis
Keywords: Olive oil; Erythrocyte membrane fatty acid contents; Oleic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stir-fried olive oil group (Experimental): olive oil in heated under 150 degrees
  Interventions: Dietary Supplement: Stir-fried olive oil group
- Natural olive oil group (Experimental): olive oil in without heated
  Interventions: Dietary Supplement: Natural olive oil group

INTERVENTIONS:
Dietary Supplement: Stir-fried olive oil group — Stir-fried olive oil group taking food with extra-virgin olive oil in stir fried food or any food with olive oil in heated under 150 degrees of celsius minimal dose per week is 30gram, providing amount of olive oil with meals is 10gram, three times in a weeks
  Arms: Stir-fried olive oil group
Dietary Supplement: Natural olive oil group — Natural olive oil group taking food with extra-virgin any food with olive oil in , minimal dose per week is 30grams, providing amount of olive oil with meals is 10gram, three times in a weeks
  Arms: Natural olive oil group

SUMMARY:
Patients with chronic kidney disease (CKD) have higher mortality rate than general population. Especially, the most common cause of mortality was known as cardiovascular disease that account for almost 50 percent in patients with dialysis. Mediterranean diet was reported for lowering risk of coronary artery disease in general population. Mediterranean diet is not acceptable in CKD patients because of restriction of potassium, phosphorus, and protein.

Relatively proper food among Mediterranean diet for hemodialysis patients is olive oil. Many researchers usually preferred olive oil as control group for evaluating effect of omega-3 fatty acid. However, previous studies reported that control groups using olive oil of 3g in a day have shown increased components of omega-3 fatty acid such as eicosapentaenoic acid (EPA) or docosahexaenoic acid (DHA). Therefore, cardioprotective effect of olive oil may be associated with increasing of omega-3 fatty acid levels.

DETAILED DESCRIPTION:
Fatty acid contents of erythrocyte membrane as a biomarker that reveals status of fatty acid within recent 3 months. Omega-3 fatty acid such as EPA or DHA, omega-3 index that calculated by sum of EPA and DHA, and ratio of EPA/arachidonic aicd (AA) are frequently reported as important biomarkers of its association with cardiovascular accidents. One of the fatty acid contents of erythrocyte membrane, oleic acid was increased in patients with acute coronary disease compared to control group. Oleic acid of erythrocyte membrane in hemodialysis patients with taking omega-3 was significantly decreased compared to group with taking olive oil. In addition, control group using olive oil was also meaningfully decreased erythrocyte membrane oleic acid compared to baseline levels. In this way, olive oil seemed to have similar effect as omega-3 fatty acid. supplement of enough amount olive oil with balanced meal may show similar effect of omega-3 fatty acid supplementation.

It is ideal way to intake olive oil in uncooked state with vegetables or breads, but practically peoples stir-fry or fry foods in olive oil instead of cooking oil. Ignition point of olive oil is 185-205 degrees of Celsius with depending on its oxidation degrees. There is a study that the contents of vitamin C in broccoli were scantly changed when broccoli was stir-fried in olive oil. It needs to identify the change of erythrocyte membrane contents between taking uncooked or natural olive oil and taking fried or stir fried olive oil with other foods. Taking meals with olive oil can change erythrocyte membrane fatty acid contents including oleic acid in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Over 20 years and under 80 years , men and women who are undergoing hemodialysis at least 6months
* Agree to participate in the clinical trial

Exclusion Criteria:

* Use of omega-3 fatty acid currently or within 3 months
* Intake over 10 gram of olive oil three times a week within 3 months
* Admitted to the hospital with cardiovascular or infectious disease within 3months
* Pregnant or expected to be pregnant
* Accompanied Liver cirrhosis or malignant tumor
* Serum albumin < 3.0 g/dL at the time of inclusion

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Erythrocyte membrane including oleic acid | 3 months after intervention
  Difference between before taking olive oil and 3 month after about erythrocyte membrane including oleic acid in patient with hemodialysis

SECONDARY OUTCOMES:
Total cholesterol | 3months after intervention
  Difference between before taking olive oil and 3 month after about total cholesterol
triglyceride | 3months after intervention
  Difference between before taking olive oil and 3 month after about triglyceride
LDL-cholesterol | 3months after intervention
  Difference between before taking olive oil and 3 month after about LDL-cholesterol
HDL-cholesterol | 3months after intervention
  Difference between before taking olive oil and 3 month after about HDL-cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: WON SUK AN, Principal Investigator — Dong-A University
Locations (1):
- Dong-A University, Busan, Seogu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Foley RN. Clinical epidemiology of cardiovascular disease in chronic kidney disease. J Ren Care. 2010 May;36 Suppl 1:4-8. doi: 10.1111/j.1755-6686.2010.00171.x. PMID 20586894
- [Background] Keith DS, Nichols GA, Gullion CM, Brown JB, Smith DH. Longitudinal follow-up and outcomes among a population with chronic kidney disease in a large managed care organization. Arch Intern Med. 2004 Mar 22;164(6):659-63. doi: 10.1001/archinte.164.6.659. PMID 15037495
- [Background] Keys A, Menotti A, Karvonen MJ, Aravanis C, Blackburn H, Buzina R, Djordjevic BS, Dontas AS, Fidanza F, Keys MH, et al. The diet and 15-year death rate in the seven countries study. Am J Epidemiol. 1986 Dec;124(6):903-15. doi: 10.1093/oxfordjournals.aje.a114480. PMID 3776973
- [Background] Martinez-Gonzalez MA, Salas-Salvado J, Estruch R, Corella D, Fito M, Ros E; PREDIMED INVESTIGATORS. Benefits of the Mediterranean Diet: Insights From the PREDIMED Study. Prog Cardiovasc Dis. 2015 Jul-Aug;58(1):50-60. doi: 10.1016/j.pcad.2015.04.003. Epub 2015 May 1. PMID 25940230
- [Background] Lee SM, Son YK, Kim SE, An WS. The effects of omega-3 fatty acid on vitamin D activation in hemodialysis patients: a pilot study. Mar Drugs. 2015 Jan 28;13(2):741-55. doi: 10.3390/md13020741. PMID 25636157
- [Background] Lee SM, Chung SH, Park Y, Park MK, Son YK, Kim SE, An WS. Effect of Omega-3 Fatty Acid on the Fatty Acid Content of the Erythrocyte Membrane and Proteinuria in Patients with Diabetic Nephropathy. Int J Endocrinol. 2015;2015:208121. doi: 10.1155/2015/208121. Epub 2015 May 18. PMID 26089878
- [Background] An WS, Lee SM, Son YK, Kim SE, Kim KH, Han JY, Bae HR, Park Y. Effect of omega-3 fatty acids on the modification of erythrocyte membrane fatty acid content including oleic acid in peritoneal dialysis patients. Prostaglandins Leukot Essent Fatty Acids. 2012 Jan-Feb;86(1-2):29-34. doi: 10.1016/j.plefa.2011.10.009. Epub 2011 Nov 8. PMID 22071008
- [Background] An WS, Lee SM, Son YK, Kim SE, Kim KH, Han JY, Bae HR, Rha SH, Park Y. Omega-3 fatty acid supplementation increases 1,25-dihydroxyvitamin D and fetuin-A levels in dialysis patients. Nutr Res. 2012 Jul;32(7):495-502. doi: 10.1016/j.nutres.2012.06.005. Epub 2012 Jul 20. PMID 22901557
- [Background] Leaf A, Kang JX, Xiao YF, Billman GE. Clinical prevention of sudden cardiac death by n-3 polyunsaturated fatty acids and mechanism of prevention of arrhythmias by n-3 fish oils. Circulation. 2003 Jun 3;107(21):2646-52. doi: 10.1161/01.CIR.0000069566.78305.33. No abstract available. PMID 12782616
- [Background] Harris WS, Von Schacky C. The Omega-3 Index: a new risk factor for death from coronary heart disease? Prev Med. 2004 Jul;39(1):212-20. doi: 10.1016/j.ypmed.2004.02.030. PMID 15208005
- [Background] Block RC, Harris WS, Reid KJ, Spertus JA. Omega-6 and trans fatty acids in blood cell membranes: a risk factor for acute coronary syndromes? Am Heart J. 2008 Dec;156(6):1117-23. doi: 10.1016/j.ahj.2008.07.014. Epub 2008 Oct 14. PMID 19033007
- [Background] An WS, Kim SE, Kim KH, Lee S, Park Y, Kim HJ, Vaziri ND. Comparison of fatty acid contents of erythrocyte membrane in hemodialysis and peritoneal dialysis patients. J Ren Nutr. 2009 Jul;19(4):267-74. doi: 10.1053/j.jrn.2009.01.027. PMID 19539181
- [Background] Moreno DA, Lopez-Berenguer C, Garcia-Viguera C. Effects of stir-fry cooking with different edible oils on the phytochemical composition of broccoli. J Food Sci. 2007 Jan;72(1):S064-8. doi: 10.1111/j.1750-3841.2006.00213.x. PMID 17995900